CLINICAL TRIAL: NCT04346017
Title: Evaluation of Interleukine 6 (and Other Cytokines and Inflammatory Markers) in SARS-Cov-2 Infected Patients With a Systemic Inflammatory Response Syndrome
Brief Title: Evaluation of Interleukine 6 (and Other Cytokines and Inflammatory Markers) in COVID-19 Patients With a Systemic Inflammatory Response Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Corazza (Other)
Responsible Party: Sponsor-Investigator, Francis Corazza, Head of the Immunology Laboratory, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-IL6-COVID-19
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilation support (Experimental): The experimental group will include Covid-19 infected patients with non-invasive or invasive ventilation support (BCRSS score ≥3).
  Interventions: Diagnostic Test: Cytokines dosage; Diagnostic Test: Complement dosage
- Control group (Other): The control group will include Covid-19 infected patients who don't have respiratory problems justifying a transfer to intensive care.
  Interventions: Diagnostic Test: Cytokines dosage; Diagnostic Test: Complement dosage

INTERVENTIONS:
Diagnostic Test: Cytokines dosage — Dosage of inflammatory cytokines and other markers of systemic inflammatory syndromes (TNFa, IFNg, IL1, IL7, IL10, IL12, IL17, sCD25, sCD163, sCD14, IL-6, IL6-R, complex IL6-IL6R, glycolsylated ferritin...).
Diagnostic Test: Complement dosage — Dosage of the complement parameters: CH50, C3, C4, C3d, C5a, SC5b-9, C4a, MASP-2.

SUMMARY:
In patients infected by the SARS-Cov-2 Coronavirus a severely progressive disease requiring hospitalization in intensive care seems related to deregulation of cytokines with very high levels of IL-6, IL-2, IL-7, IL-10 and TNF-α. In order to elucidate the mechanism of this hyper inflammatory syndrome we will measure a panel of pro and anti inflammatory cytokines, as well as known markers of macrophage activation syndrome.

To determine the role of activation of the complement cascade the most important complement factors and their activation markers will be measured.

The changes of those parameters will be monitored after administration of an anti-IL6R antibody therapy.

DETAILED DESCRIPTION:
In patients with severely progressive SARS-Cov-2 Coronavirus infection, the elderly and immunocompromised are at greater risk of progressing to a serious image of ARDS (Acute Respiratory Distress syndrome). A recent study has shown that patients, sometimes young, requiring hospitalization in intensive care have deregulation of cytokines with very high levels of IL-6, IL-2, IL-7, IL-10 and TNF-α. The cytokines involved in the pathogenesis and clinical manifestations of CRS are mainly IL-6, gamma interferon (IFN-g), tumor necrosis factor alpha (TNF-a) and IL-10.

Although immunoinflammatory therapy is not systematically recommended in pneumonia linked to SARS-CoV-2, given the CRS and the pathophysiological results of pulmonary edema and the formation of the hyaline membrane, a targeted therapeutic approach and temporally accompanied by adequate ventilatory support could be beneficial in patients with severe pneumonia who develop ARDS. Tocilizumab (Roactemra®) is a drug that blocks the IL-6 receptor commonly prescribed for the treatment of rheumatoid arthritis. The intravenous formulation has been approved for the treatment of CRS which occurs during treatment with Car-T; given the clinical picture and cytokine levels in patients with severe SARS-Cov-2 pneumonia, Tocilizumab or another anti-IL6R antagonist may reasonably be expected to contribute to the control of virus-induced Systemic Inflammatory Response Syndrome (SIRS) in patients with elevated levels of IL-6.

The objectivation of high interleukin 6 levels in these patients should be an important scientific argument to justify the administration of therapy based on antagonization of IL6. Measurement of other pro inflammatory cytokines will shed light on the mechanism of the inflammatory syndrome induced by the SARS-CoV-2 virus.

One of the pathophysiological mechanisms of pulmonary pathology could be the induction of the production of complement factors by interleukin 6 as well as the activation of the complement cascade by the virus via the lectin pathway. It is known that one of the effects of Tocilizumab is to reduce the concentration of the various complement factors, the synthesis of which is under the control of interleukin 6. This is why this study proposes to measure certain parameters of the complement (CH50, C3, C4, C3d, C5a, SC5b-9, C4a, MASP-2) in order to objectify and quantify this activation.

If the activation of the complement proves significant it could be an argument for a treatment targeting more specifically the cascade of the complement.

ELIGIBILITY:
Inclusion Criteria:

* End of the initial phase of high viral load of SARS-Cov-2 (for example apyretic> 72h and / or at least 7 days after the onset of symptoms)
* Worsening of respiratory exchanges which require non-invasive or invasive ventilation support (BCRSS score ≥3)
* High levels of IL-6 (> 40 pg / ml); alternatively high levels of d-dimer and / or PCR and / or ferritin and / or fibrinogen gradually increase.
* A control group will be formed by patients in the Covid unit who do not have respiratory problems justifying a transfer to intensive care.

Exclusion Criteria:

* Documented sepsis caused by other pathogens other than SARS-Corv-2.
* Presence of comorbidities likely to lead, according to clinical judgment, to an unfavorable result
* Immunosuppressive anti-rejection therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
IL6 concentration | Before anti-IL6R treatment (baseline)
  Interleukine 6, soluble IL6-R, complex IL6-IL6R concentration
IL6 concentration change from baseline value | Twice a week from day 1 to day 14 post anti-IL6R administration
  Interleukine 6 soluble IL6-R, complex IL6-IL6R variation compared to baseline value
Complement parameters | Before anti-IL6R treatment (baseline)
  CH50, C3, C4, C3d, C5a, SC5b-9, C4a, MASP-2
Complement parameters change from baseline values | Twice a week from day 1 to day 14 post anti-IL6R administration
  CH50, C3, C4, C3d, C5a, SC5b-9, C4a, MASP-2 variation compared to baseline values
Inflammatory cytokines baseline concentrations | Before anti-IL6R treatment (baseline)
  Concentration of TNFa, IFNg, IL1, IL7, IL10, IL12, IL17, IL18
Inflammatory cytokines change from baseline values | Twice a week from day 1 to day 14 post anti-IL6R administration
  Concentration of TNFa, IFNg, IL1, IL7, IL10, IL12, IL17, IL18 variation compared to baseline values

SECONDARY OUTCOMES:
Concentration of markers of macrophage activation | Before anti-IL6R treatment (baseline)
  sCD25, sCD163, sCD14, glycosylated ferritin
Markers of macrophage activation change from baseline values | Twice a week from day 1 to day 14 post anti-IL6R administration
  sCD25, sCD163, sCD14, glycosylated ferritin variation compared to baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ponthieux F, Dauby N, Maillart E, Fils JF, Smet J, Claus M, Besse-Hammer T, Bels D, Corazza F, Nagant C. Tocilizumab-Induced Unexpected Increase of Several Inflammatory Cytokines in Critically Ill COVID-19 Patients: The Anti-Inflammatory Side of IL-6. Viral Immunol. 2022 Jan-Feb;35(1):60-70. doi: 10.1089/vim.2021.0111. Epub 2022 Jan 27. PMID 35085462